CLINICAL TRIAL: NCT04531306
Title: An Analysis of Kinesio® Tape on Myofascial Pain Syndrome of the Iliotibial Band
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Dakota State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HE20151
Record Dates: First submitted 2020-05-21; First posted 2020-08-28 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Myofascial Trigger Point Pain
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pre-tape (Active Comparator)
  Interventions: Other: Kinesio® Tape
- With tape 1 (Experimental)
  Interventions: Other: Kinesio® Tape
- With tape 2 (Experimental)
  Interventions: Other: Kinesio® Tape
- Post-tape (Experimental)
  Interventions: Other: Kinesio® Tape

INTERVENTIONS:
Other: Kinesio® Tape — Fascial taping technique for myofascial trigger points on the iliotibial band

SUMMARY:
Participants will report for two research sessions. Prior to arrival, membership to a club sports team will be confirmed via email. The first session will require one hour, while the second will require 30 minutes. Maximum amount of time expected is one and a half hours, over two sessions in 48 hours. The 1st and 2nd sessions will be separated by 48 hours. Upon arrival for session 1, informed consent will be obtained along with the following demographic information: age, sex, height, weight, dominant leg, and sport. Next, the participant will complete the Musculoskeletal Questionnaire (MQ) in regard to the last 12 months. Participants will then be assessed for trigger points in their dominant side iliotibial band via palpation. Diagnostic criteria for trigger point will be modeled after Travell and Simons: taut band, pain upon palpation, referred pain, and a local twitch response. Up to four trigger points will be marked on the subject's skin with marker or pen. Pain pressure threshold will be obtained via algometer, using the terminology "Tell me the first moment you experience pain by verbalizing 'pain' ". Then, three pain pressure threshold readings will be taken per trigger point and then averaged by the researcher. Kinesiology tape will then be applied to the identified trigger points using the Fascial Technique. Pain pressure threshold will be obtained again with the same protocols 10 minutes after the tape is applied. The participant will be asked to wear the tape for 48 hours. Upon arrival for session 2, the application of the tape will be confirmed. With the participant's choice to continue in the study, a third and fourth measurement of pain pressure threshold will be obtained: one with the tape remaining on, and another 10 minutes after removal of the tape. Again, three pain pressure threshold readings will be taken per trigger point and then averaged by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* member of club sports team

Exclusion Criteria:

* acute quadriceps strain in last six months
* knee surgery in last six months
* acute hamstring strain in last six months
* allergy to adhesive
* malignancies
* cellulitis
* skin infection
* diabetes
* fragile skin

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-10-04 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
with-in subject differences pre- and 10-minute post- tape application | 10 minutes
  measured by pain pressure threshold (N/s2) via algometer
with-in subject differences pre- and 48-hour post- tape application | 48 hours
  measured by pain pressure threshold (N/s2) via algometer
with-in subject differences 10-minute post- and 48-hour post- tape application | 48 hours
  measured by pain pressure threshold (N/s2) via algometer
with-in subject differences 48-hour post- tape application and post- 10- minute tape removal | 10 minutes
  measured by pain pressure threshold (N/s2) via algometer

CONTACTS AND LOCATIONS:
Locations (1):
- North Dakota State University, Fargo, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No